CLINICAL TRIAL: NCT01363375
Title: The Investigation of Biomechanical Mechanism of Different Foot Structures on Plantar Fasciitis and the Evaluation of Efficacy on Therapeutic Footwear
Brief Title: Effects of Different Foot Structures on Plantar Fasciitis and Therapeutic Footwear Intervention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chih-Chin Hsu, Department of physical medicine and rehabilitation, Chang Gung Memorial Hospital at Keelung
Other Study IDs: NSC 97-2320-B-027-002-MY3
Record Dates: First submitted 2011-05-10; First posted 2011-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2008-02

CONDITIONS: Fasciitis
Keywords: Plantar fascia; Plantar fasciitis; Foot orthosis; Finite element analysis; Gait analysis; Plantar pressure measurement
MeSH Terms: conditions — Fasciitis; Fasciitis, Plantar | interventions — Foot Orthoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- normal foot: Subjects with normal foot structure
  Interventions: Procedure: Foot orthosis, footwear
- flat foot: Subjects with flat foot structure.
  Interventions: Procedure: Foot orthosis, Footwear
- high arch foot: Subjects with high arch foot structure.
  Interventions: Procedure: Foot orthosis, footwear

INTERVENTIONS:
Procedure: Foot orthosis, footwear — flat insole, total contact insole , carbon fiber plate; general shoe and rocker sole shoe
  Other Names: Carbon fiber enhancement; Rocker sole shoe
  Groups: normal foot
Procedure: Foot orthosis, Footwear — flat insole, total contact insole, carbon fiber plate; general shoe and rocker sole shoe
  Other Names: Carbon fiber enhancement; Rocker sole shoe
  Groups: flat foot
Procedure: Foot orthosis, footwear — flat insole, total contact insole, carbon fiber plate; general shoe and rocker sole shoe
  Other Names: Carbon fiber enhancement; Rocker sole shoe
  Groups: high arch foot

SUMMARY:
Excessive repetitive loading concentrating upon plantar fascia is considered as the most influential factor in plantar fasciitis development. Abnormal foot structure may lead to high risk of plantar fasciitis. However, the biomechanical factor that may cause plantar fasciitis has not been thoroughly investigated. Orthotic device is a common treatment used for plantar fasciitis. However, there is no direct and quantitative data, such as stress and strain distribution of plantar fascia for patient with foot orthosis during gait. Therefore, the aim of this three-year project study is to investigate the biomechanical mechanism of different foot structures and to understand the biomechanical response of plantar fascia during stance phase of gait cycle by dynamic finite element analysis, gait analysis as well as plantar pressure measurement. In addition, the efficacy of foot orthoses will be evaluated by the same research process. The hypotheses are that flat foot and high arch foot may result in higher stress and strain upon plantar fascia during gait; the foot orthosis, such as total contact insole, carbon fiber plate and rocker bottom sole, would reduce stress and strain distribution around the calcaneal medial tuberosity; rigid and curved geometric bottom will be able to relief plantar fascia stretching during push-off phase.

DETAILED DESCRIPTION:
The plantar fascia has long been considered to play an important role in the weight-bearing foot, both in static stance and in dynamic function. Various functional and structural roles have been indicated by virtue of its anatomical attachments. Excessive repetitive loading concentrating upon plantar fascia is considered as the most influential factor in plantar fasciitis development. Abnormal foot structure may lead to high risk of plantar fasciitis. However, the biomechanical factor that may cause plantar fasciitis has not been thoroughly investigated. Orthotic device is a common treatment used for plantar fasciitis. However, there is no direct and quantitative data, such as stress and strain distribution of plantar fascia for patient with foot orthosis during gait. Therefore, the aim of this three-year project study is to investigate the biomechanical mechanism of different foot structures and to understand the biomechanical response of plantar fascia during stance phase of gait cycle by dynamic finite element analysis, gait analysis as well as plantar pressure measurement. In addition, the efficacy of foot orthoses will be evaluated by the same research process.

In this research, a plantar fascia specific finite element foot model with tibia will be reconstructed from magnetic resonance images obtained from subjects with normal foot, flat foot and high arch foot structures. The same subject will also serve for plantar soft tissue material property testing, gait analysis as well as plantar pressure measurement. The kinematic and kinetic data from both gait analysis and plantar pressure measurement will be used to validate the accuracy of dynamic finite element analysis. In addition, 20 normal, 10 flat foot and 10 high-arch foot subjects will also be recruited for gait analysis and plantar pressure measurement. The kinematic and kinetic data from both gait analysis and plantar pressure measurement will be compared with the results of finite element analysis.

ELIGIBILITY:
Inclusion Criteria:

1. With normal bilateral foot arch structure, unilateral flat foot or unilateral high arch foot
2. With no more musculoskeletal disorders or malalignment
3. With no degeneration of low-extremity joint
4. With no diabetes mellitus or peripheral neuropathy
5. With no injury and pain of low-extremity in recent three month.

Exclusion Criteria:

1. Painful disorders
2. Foot related disorders or deformity
3. Dorsal or plantar wound and trauma
4. Poor proprioception
5. Obvious abnormal gait pattern, such as midfoot strike

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with normal foot structure or abnormal foot structure (flat foot or high arch foot) will be invited to participant this study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Gait parameter, plantar pressure. | 1 day
  Gait parameter, such as MTP joint range of motion(degree), meidal longitudinal arch angle(degree), hindfoot eversion/inversion angle(degree).
  Plantar pressure, such as peak pressure(kPa), center of pressure trajectory(mm/s).

SECONDARY OUTCOMES:
Foot MRI image, foot plantar soft tissue material property. | 1 day
  Foot plantar soft tissue material property, such as elastic modulus(N/mm^2).

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chin Hsu, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital, Keelung
Locations (1):
- Chang Gung Memorial Hospital@ Taoyuan, Taoyuan District, Taiwan, Taiwan

REFERENCES:
- [Background] Boyer KA, Andriacchi TP. Changes in running kinematics and kinetics in response to a rockered shoe intervention. Clin Biomech (Bristol). 2009 Dec;24(10):872-6. doi: 10.1016/j.clinbiomech.2009.08.003. Epub 2009 Sep 9. PMID 19744753
- [Background] Van Bogart JJ, Long JT, Klein JP, Wertsch JJ, Janisse DJ, Harris GF. Effects of the toe-only rocker on gait kinematics and kinetics in able-bodied persons. IEEE Trans Neural Syst Rehabil Eng. 2005 Dec;13(4):542-50. doi: 10.1109/TNSRE.2005.858460. PMID 16425836
- [Background] Brown D, Wertsch JJ, Harris GF, Klein J, Janisse D. Effect of rocker soles on plantar pressures. Arch Phys Med Rehabil. 2004 Jan;85(1):81-6. doi: 10.1016/s0003-9993(03)00374-5. PMID 14970973
- [Background] Caravaggi P, Pataky T, Gunther M, Savage R, Crompton R. Dynamics of longitudinal arch support in relation to walking speed: contribution of the plantar aponeurosis. J Anat. 2010 Sep;217(3):254-61. doi: 10.1111/j.1469-7580.2010.01261.x. Epub 2010 Jul 14. PMID 20646107
- [Background] Caravaggi P, Pataky T, Goulermas JY, Savage R, Crompton R. A dynamic model of the windlass mechanism of the foot: evidence for early stance phase preloading of the plantar aponeurosis. J Exp Biol. 2009 Aug;212(Pt 15):2491-9. doi: 10.1242/jeb.025767. PMID 19617443
- [Derived] Lin SC, Chen CP, Tang SF, Wong AM, Hsieh JH, Chen WP. Changes in windlass effect in response to different shoe and insole designs during walking. Gait Posture. 2013 Feb;37(2):235-41. doi: 10.1016/j.gaitpost.2012.07.010. Epub 2012 Aug 9. PMID 22884544